CLINICAL TRIAL: NCT02811744
Title: 11C-Acetate Position Emission Tomography/Computerized Tomography (PET/CT) Imaging As a Biomarker of Amyloid-Induced Neuroinflammation
Brief Title: 11C-Acetate PET/CT Imaging As a Biomarker of Amyloid-Induced Neuroinflammation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding issues.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 824822
Record Dates: First submitted 2016-06-20; First posted 2016-06-23 (Estimated); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — carbon-11 acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amnestic MCI cohort (Experimental): Patients with Mild Cognitive Impairment (MCI) (up to 14) will be recruited primarily from the Penn Memory Center (PMC). Clinical diagnostic criteria (described in further detail in Study Procedures section) will be used to identify subjects who are meet criteria for amnestic MCI. Participants will receive injection of radioactive tracer 11C-acetate and complete a PET/CT scan.
  Interventions: Drug: 11C-acetate
- Control cohort (Other): Normal control subjects in the same age range (up to 6) will be recruited from a current ongoing study investigating neuroinflammation in late life depression and healthy controls, from the control group in which all subjects receive MRI and lumbar puncture (LP) and from the PMC research cohort. Participants will receive injection of radioactive tracer 11C-acetate and complete a PET/CT scan.
  Interventions: Drug: 11C-acetate

INTERVENTIONS:
Drug: 11C-acetate — Participants will receive injection of radioactive tracer 11C-acetate and complete a PET/CT scan.

SUMMARY:
The proposed study aims to use 11C-acetate position emission tomography/computed tomography (PET/CT) to preliminarily test and validate methods for imaging astrocyte activation as an early indicator of neuroinflammation in Alzheimer's disease (AD). 11C-Acetate PET/CT has been shown to quantify astrocyte activation in vivo, but no reports have evaluated its potential in AD. The investigators propose to test 11C-Acetate PET/CT as a marker for astrocyte activation associated with pathologic amyloid deposition in AD. The investigators will compare binding between subjects with early stage AD and healthy controls. Further, the investigators will investigate the correlation between amyloid and acetate binding. If the investigators find increased astrocyte activation in response to cerebral amyloid by showing a group difference in brain acetate uptake between disease and controls or a strong correlation between acetate and amyloid PET/CT binding. Validating neuroinflammation markers in AD ultimately may guide therapeutic modulation of beneficial and damaging neuroinflammation to slow disease progression, as well as providing new insights into AD pathophysiology.

ELIGIBILITY:
Inclusion Criteria for amnestic MCI cohort:

1. Participants will be at least 65 years of age
2. Positive brain amyloid PET/CT scan within 6 months of study screening
3. Mini-mental status examination (MMSE) score ≥ 24 at screening visit
4. A brain MRI is required. If a brain MRI has been performed within 6 months of 11C-Acetate PET/CT and of adequate quality that scan may be used for the study analysis, subjects who do not have a brain MRI will undergo a brain MRI as a part of this study
5. Participants must identify a study partner who is willing to accompany the patient to study visits
6. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures. If the patient is unable to provide informed consent, the patient's legal representative may consent on behalf of the patient but the patient will be asked to confirm assent.

Inclusion Criteria for Control cohort:

1. Participants will be at least 65 years of age
2. History of negative brain amyloid PET/CT scan within 6 months of study screening OR negative cerebrospinal fluid (CSF) analysis for AD biomarkers within 6 months of study screening
3. Mini-mental status examination (MMSE) > 27 at screening visit
4. A brain MRI is required. If a brain MRI has been performed within 6 months of enrollment to this study and of adequate quality that scan may be used for the study analysis, subjects who do not have a brain MRI will undergo a brain MRI as a part of this study
5. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria for both cohorts:

1. Inability to tolerate or contraindication to imaging procedures (PET/CT or MRI) in the opinion of an investigator or treating physician
2. History of stroke or other neurological disease that in the opinion of the investigator might interfere with evaluation of the 11C-Acetate scan
3. Any medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Nasrallah, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 MCI subjects and 5 Healthy Controls recruited from neurology practice at University of Pennsylvania
Pre-assignment Details: 11 subjects were enrolled. Target enrollment of 20 was not met due to difficulty with recruitment.
Groups:
- Control Cohort: Normal control subjects in the same age range (up to 6) will be recruited from a current ongoing study investigating neuroinflammation in late life depression and healthy controls, from the control group in which all subjects receive MRI and LP and from the PMC research cohort. Participants will receive injection of radioactive tracer 11C-acetate and complete a PET/CT scan.
  11C-acetate: Participants will receive injection of radioactive tracer 11C-acetate and complete a PET/CT scan.
Period: Overall Study
Arm/Group | Amnestic MCI Cohort | Control Cohort
Started | 6 | 5
Completed | 6 (6 MCI patients were enrolled and completed the PET/CT scan) | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amnestic MCI Cohort | Control Cohort | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 3 | 8
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 11C-acetate Uptake in Amyloid Positive Mild Cognitive Impairment (MCI) Subjects Versus Amyloid Negative Healthy Controls
Description: We compare the whole brain 11C-acetate uptake standardized uptake value ratio (SUVR) between the amnestic MCI and control cohorts. Static summed images from 40-60 minutes after tracer injection were generated from raw dynamic PET data. This timeframe was selected to preferentially capture 11C-acetate trapped in biosynthetic pathways in activated astrocytes, rather than what was catabolized to 11C-CO2 .Mean tracer binding, expressed as standardized uptake values (SUV) in the whole cerebral cortex and other regions is measured from these summed images using PMOD software (PMOD technologies). SUVR is generated by dividing the mean whole cortex SUV by the mean cerebellar gray matter SUV; SUVR is a unitless measure. For this tracer, higher values are worse, indicating more astrocyte activation and inflammation.
Time Frame: 6 months
Population: There were six participants with MCI and 2 controls
Measure: Mean (Standard Deviation); unit: Standardized uptake value ratio (SUVR)
Arm/Group | Amnestic MCI Cohort | Control Cohort
Number analyzed (Participants) | 6 | 2
Standardized uptake value ratio (SUVR) | 1.04 (0.06) | 1.04 (0.05)
Statistical Analysis 1: Comparison: Amnestic MCI Cohort vs Control Cohort; No power calculation. This is an exploratory study; Test type: Equivalence — Equivalence was defined as no significant difference between study groups on a T-test; p = 0.5, t-test, 2 sided — No adjustments on the comparison. There was no multiple comparison adjustment for the p value, as this was the primary outcome. This is the experimental p value; the threshold for significance was 0.05

ADVERSE EVENTS:
Time Frame: 24 hours post 11C-Acetate injection
Description: No adverse events reported
Arm/Group | Amnestic MCI Cohort | Control Cohort
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT02811744/Prot_SAP_000.pdf